CLINICAL TRIAL: NCT05828927
Title: enCompass Carolina: A Social Support and Coaching Program for Cancer Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: The Duke Endowment (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2242
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: social support; rural; caregivers; coaching
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregiver of subject with cancer (Other): Adults who identify as a primary unpaid caregiver for a rural-dwelling adult with cancer.
  Interventions: Behavioral: Eco-mapping tool; Behavioral: Caregiver-coach study visits
- Subject with Cancer (No Intervention): Subjects is with cancer and receive care from caregivers.

INTERVENTIONS:
Behavioral: Eco-mapping tool — The web application allows caregivers to visually identify and organize their existing social network (family, friends, community of worship, and others) to assist with their support needs, tailored to their context. For each of the six support social support domains (in-home, informational, communication, financial, emotional and spiritual, transportation (e.g., emotional, informational, practical), the enCompass web application prompts the individual to identify members of their network. After completing each domain, caregivers are presented with a visual social support
  Arms: Caregiver of subject with cancer
Behavioral: Caregiver-coach study visits — Caregivers engage in up to 8 manualized, telephone/videoconference visits with a trained caregiver coach. The caregiver coach uses the study manual and interview guide to provide support for caregiver support-seeking and problem-solving.
  Arms: Caregiver of subject with cancer

SUMMARY:
This study explores the feasibility, acceptability, and preliminary efficacy of a social support intervention in cancer caregivers who live in rural communities. Cancer caregivers need support, especially when they live at a distance from healthcare centers. enCompass Carolina is a social support intervention, that supports caregivers by helping them find and use new sources of support. The purpose of this study is to test and receive feedback about the program.

ELIGIBILITY:
Inclusion Criteria

Inclusion criteria for caregivers In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

1. English-speaking.
2. Ability to provide written or electronic informed consent to participate in the study.
3. Subject is willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.
4. Age ≥ 18 years at the time of consent. Identify as an informal (unpaid) caregiver for a rural-dwelling adult with a stage II-IV solid tumor or any hematologic malignancy in active treatment (see eligibility criteria for patients).

Inclusion criteria for subjects with cancer In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

1. Their identified caregiver is enrolled in the study
2. English-speaking.
3. Ability to provide written or electronic informed consent to participate in the study.
4. Subjects are willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.
5. Age ≥ 18 years at the time of consent. Have a diagnosis of stage II-IV solid tumor or any hematologic malignancy receiving active treatment s, not including hormonal therapy

7. Live in a rural area according to the USDA's Rural/Urban Commuting Area (RUCA) score of >4.

Exclusion Criteria

Exclusion criteria for caregivers

1. Unable to complete self-report instruments due to illiteracy, neurologic illness, inability to speak or read English, or other causes;
2. Existence of another co-morbid disease, which in the opinion of the investigator, prohibits participation in the protocol;
3. Participation in the intervention development phase of this intervention.

Exclusion criteria for subjects with cancer

1. Unable to complete self-report instruments due to illiteracy, neurologic illness, inability to speak or read English, or other causes;
2. Existence of another co-morbid disease, which in the opinion of the investigator, prohibits participation in the protocol;
3. Their caregiver does not enroll in the study or withdraws consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Study feasibility - caregiver enrollment | 8 weeks
  Study feasibility will be measured by caregiver enrollment rates, defined as the proportion of eligible caregivers approached about the study who consent to participate.
Study feasibility - Caregiver intervention engagement | 8 weeks
  Study feasibility will be measured by caregiver intervention engagement, defined as the proportion of enrolled caregiver subjects who receive at least one intervention visit.

SECONDARY OUTCOMES:
Intervention acceptability-qualitative | 4 weeks, 8 weeks
  Intervention acceptability will be measured using the Acceptability of the Intervention Measure (AIM) survey scores.
  AIM is a survey questionnaire that includes 4 questions. Response Scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree. Scoring Instructions: Scales can be created for each measure by averaging responses. Scale values range from 1 to 5. No items need to be reverse-coded.
Intervention acceptability-quantitative | 4 weeks, 8 weeks
  Intervention acceptability will be evaluated using thematic analysis of post-intervention semi-structured interviews.
Caregiver self-efficacy | Baseline, 4 weeks, 8 weeks
  Caregiver self-efficacy will be measured using the Coping Self-Efficacy Scale (CSES).
  The CSES is a 26-item measure of one's confidence in performing coping behaviour when facing life challenges. It measures the use of problem-focused coping, receiving of social support and stopping unpleasant emotions and thoughts. Scores range from not at all confident=0 to very confident=100. A score of 0 means 'extremely low self efficacy' and a score of 100 means 'extremely high self efficacy'.

CONTACTS AND LOCATIONS:
Overall Officials: Erin E Kent, PhD, MS, Principal Investigator — Department of Health Policy and Management Gillings School of Global Public Health
Locations (1):
- UNC Lineberger, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Kent EE, Tan KR, Nakamura ZM, Kovacs J, Gellin M, Deal A, Park EM, Reblin M. Building on and tailoring to: Adapting a cancer caregiver psychoeducational intervention for rural settings. Cancer Med. 2024 Sep;13(17):e70187. doi: 10.1002/cam4.70187. PMID 39234997